CLINICAL TRIAL: NCT05008575
Title: Phase I Study to Evaluate the Safety and Effectiveness of Anti-CD33 CAR NK Cell Therapy in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Anti-CD33 CAR NK Cells in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xi Zhang, MD, chef of hemotology department, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD33 CAR NK-AML
Record Dates: First submitted 2021-08-14; First posted 2021-08-17 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- antiCD33 CAR NK cells (Experimental): After preconditioning with chemotherapy, the antiCD33 CAR NK cells will be evaluated
  Interventions: Biological: anti-CD33 CAR NK cells; Drug: Fludarabine; Drug: Cytoxan

INTERVENTIONS:
Biological: anti-CD33 CAR NK cells — 6×10^8, 12×10^8, 18×10^8/KG Treatment follows a lymphodepletion
Drug: Fludarabine — recommendation: 30mg/m2 (D-5~D-3),determined by tumor burden at baseline.
Drug: Cytoxan — recommendation: 300-500mg/m2 (D-5~D-3),determined by tumor burden at baseline.

SUMMARY:
CAR technology has been used in T cell therapy and gets great success in treating hematological diseases. Following models of CAR T cells, CAR NK cell therapy has been one hot point. For myeloid malignancies, CD33 is widely expressed. Targeting CD33 surface antigens by CAR NK cells provides an off-the-shelf immune cell therapy.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status score ≤ 2.
2. Life expectancy ≥ 12 weeks from the time of enrollment.
3. Disease status at the time of enrollment: -Patients with AML (except M3) who have not achieved complete remission after standard chemotherapy regimens; -Not suitable or unconditional for allogeneic hematopoietic stem cell transplantation; -Patients with recurrent acute myeloid leukemia after autologous hematopoietic stem cell transplantation without active graft-versus-host disease (GVHD).
4. CD33 expression must be detected on greater than 50% of the malignant cells by immunohistochemistry or greater than 80% by flow cytometry.
5. Adequate main organ function as assessed by the following laboratory requirements: creatinine ≤ 2.5 × upper limit of normal, cardiac ejection fraction ≥ 40%, oxygen saturation ≥ 90%, total bilirubin ≤ 3 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, Hgb≥80g/L.
6. Without history of accepting anti-cancer therapy, including chemotherapy, radiotherapy, immunotherapy (immune suppressive drugs or corticosteroid treatment) within 4 weeks of screening.
7. Women of child-bearing age must have evidence of negative pregnancy test.
8. Subjects of reproductive potential must agree to use acceptable birth control methods within 1 year after treatment, as described in protocol.
9. After discussion by the expert group, the patient's condition was analyzed and combined with the general physical condition of the patient, the benefit of participating in the clinical trial was greater than the risk.
10. All participants must have the ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL M3): t(15;17)(q22;q12); (promyelocytic leukemia [PML]/retinoic acid receptor [RAR] alpha [a]) and variants excluded.
2. Active acute or chronic GVHD or requirement of immunosuppressant medications for GVHD within 4 weeks of enrollment.
3. Have been diagnosed with or treated other malignant tumors other than AML within 5 years before screening, except for the following conditions: participants with adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer; or received radical treatment Local prostate cancer, ductal carcinoma in situ.
4. There are serious systemic diseases: New York Heart Association (NYHA) stage III or IV congestive heart failure; cerebrovascular accident or myocardial infarction or hemodynamic instability caused by arrhythmia within 6 months before signing the informed consent; impaired cardiac function (LVEF<50%) assessed by echocardiographic scan.
5. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
6. Pregnant or lactating women.
7. Subjects with radiologically-detected CNS chloromas or CNS 3 disease (presence of ≥ 5/μL white blood cells (WBCs) in cerebral spinal fluid (CSF) and cytospin positive for blasts [in the absence of a traumatic lumbar puncture] and/or clinical signs of CNS leukemia such as a cranial nerve palsy from active disease). Subjects with adequately treated CNS leukemia are eligible.
8. Human immunodeficiency virus (HIV) seropositivity; hepatitis B surface antigen is positive or HBV DNA is higher than the detection limit of the analysis method; hepatitis C antibody is positive or HCV RNA is higher than the detection limit of the analysis method; syphilis antibody and syphilis rapid plasma reagin are positive; CMV DNA is positive.
9. Patients who suffer from allergies for any cytokines or antibodies.
10. Contraindications for fludarabine or cyclophosphamide treatment.
11. Receiving corticosteroids at >20 mg daily prednisone dose or equivalent.
12. Drug abuse and addiction.
13. History of mental disorders.
14. Other patients that researchers considered unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate (ORR) | 4 weeks after infusion
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CRi), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
incidence of participants with dose limiting toxicity (DLT) | within 4 weeks after infusion
  To characterize the safety, tolerability of Anti-CD33 CAR NK cells

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years after infusion
Overall Response Rate (ORR) | up to 2 years after infusion
Overall survival(OS) | up to 2 years after infusion

CONTACTS AND LOCATIONS:
Overall Officials: xi zhang, MD/PhD, Principal Investigator — Department of Hematology, Xinqiao Hospital
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang R, Wang X, Yan H, Tan X, Ma Y, Wang M, Han X, Liu J, Gao L, Gao L, Jing G, Zhang C, Wen Q, Zhang X. Safety and efficacy of CD33-targeted CAR-NK cell therapy for relapsed/refractory AML: preclinical evaluation and phase I trial. Exp Hematol Oncol. 2025 Jan 2;14(1):1. doi: 10.1186/s40164-024-00592-6. PMID 39748428